CLINICAL TRIAL: NCT03098082
Title: Urine Trypsinogen 2 Dipstick for the Early Detection of Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jeffrey Easler, Assistant Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1701950933
Record Dates: First submitted 2017-03-13; First posted 2017-03-31 (Actual); Results first posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Intervention Model Description: All enrolled subjects who meet study inclusion /exclusion will have the Urine Trypsinogen dip stick test
Masking Description: Cares providers, patients and study primary investigators will be blinded to 2 hour Urine Trypsinogen dip stick test results. Results will not be released or posted on subject chart.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Actim Pancreatitis Dipstick Test (Other): All enrolled subjects who meet inclusion/exclusion criteria will have the Urine Trypsinogen 2 Dipstick test done.
  Interventions: Device: Actim Pancreatitis

INTERVENTIONS:
Device: Actim Pancreatitis — Actim Pancreatitis (Medix Biochemica) is a urine trypsinogen-2 dipstick test (UTDT) that uses trypsinogen-2 as a biomarker for acute pancreatitis.

SUMMARY:
Post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP) is the most common, serious complication of ERCP. More than 500,000 ERCP procedures are performed from which 25,000 cases of PEP occur in the U.S.A. annually. PEP accounts for significant morbidity and health care expenditures. While symptoms of PEP arise immediately after ERCP, they are non-specific. Consequently, unnecessary admissions of outpatients without PEP and inadvertent discharge of outpatients with PEP from ERCP recovery are common. An accurate, confirmatory test for diagnosis of PEP immediately after ERCP is lacking. Actim Pancreatitis (Medix Biochemica) is a urine trypsinogen-2 dipstick test (UTDT) that uses trypsinogen-2 as a biomarker for acute pancreatitis. Urine Trypisinogen-2 Dipstick test (UTDT) is a simple, inexpensive test with promising preliminary data for accuracy for immediate diagnosis of PEP. Prior studies of ITDT test characteristics lack rigorous scientific design. Investigators will enroll 1825 ERCP outpatients at our institution in a prospective cohort study. A pre-ERCP UTDT test and diagnostic UTDT 2 hours after the ERCP will be performed. Patients with a positive baseline UTDT will be followed clinically as part of this study without 2 hour testing. Care providers and study primary investigators will be blinded to the 2 hour UTDT results. Baseline, intra-procedure and recovery room clinical data will be recorded. Diagnosis of PEP will be made blinded to the UTDT result. Admission status for PEP will be assessed by review of records and phone/e-mail contact 5 days and 30 days after ERCP procedure. Sensitivity and specificity of 2 hour post ERCP UTDT for the diagnosis of PEP will be calculated.

Aims: 1) To determine the test characteristics of UTDT for the diagnosis of PEP 2 hours after completion of ERCP. 2) To identify and describe patients with baseline UTDT positivity, in whom this test offers limited utility.

Specific Aims:

Primary Aim 1.1 To determine the test characteristics (sensitivity and specificity) of the UTDT for the diagnosis of PEP:

Hypotheses:

1. UTDT is a sensitive and specific test for the diagnosis of PEP for patients undergoing ERCP.
2. At a cutpoint for a negative test of <50ug/L, UTDT will be accurate at 2 hours post ERCP in patients whose baseline test is negative.

DETAILED DESCRIPTION:
Post-endoscopic retrograde cholangiopancreatography (ERCP) pancreatitis (PEP) is the most common, serious complication of ERCP. More than 500,000 ERCP procedures are performed from which 25,000 cases of PEP occur in the U.S.A. annually. PEP accounts for significant morbidity and health care expenditures. While symptoms of PEP arise immediately after ERCP, they are non-specific. Consequently, unnecessary admissions of outpatients without PEP and inadvertent discharge of outpatients with PEP from ERCP recovery are common. An accurate, confirmatory test for diagnosis of PEP immediately after ERCP is lacking. Actim Pancreatitis (Medix Biochemica) is a urine trypsinogen-2 dipstick test (UTDT) that uses trypsinogen-2 as a biomarker for acute pancreatitis. Urine Trypisinogen-2 Dipstick test (UTDT) is a simple, inexpensive test with promising preliminary data for accuracy for immediate diagnosis of PEP. Prior studies of ITDT test characteristics lack rigorous scientific design.

Proposed Study and Methods:

Investigators will enroll 1825 ERCP outpatients at our institution in a prospective cohort study. A pre-ERCP UTDT test and diagnostic UTDT 2 hours after the ERCP will be performed. Patients with a positive baseline UTDT will be followed clinically as part of this study without 2 hour testing. Care providers and study primary investigators will be blinded to the 2 hour UTDT results. Baseline, intra-procedure and recovery room clinical data will be recorded. Diagnosis of PEP will be made blinded to the UTDT result. Admission status for PEP will be assessed by review of records and phone/e-mail contact 5 days and 30 days after ERCP procedure. Sensitivity and specificity of 2 hour post ERCP UTDT for the diagnosis of PEP will be calculated.

Aims: 1) To determine the test characteristics of UTDT for the diagnosis of PEP 2 hours after completion of ERCP. 2) To identify and describe patients with baseline UTDT positivity, in whom this test offers limited utility.

Specific Aims:

Primary Aim 1.1 To determine the test characteristics (sensitivity and specificity) of the UTDT for the diagnosis of PEP:

Hypotheses:

1. UTDT is a sensitive and specific test for the diagnosis of PEP for patients undergoing ERCP.
2. At a cutpoint for a negative test of <50ug/L, UTDT will be accurate at 2 hours post ERCP in patients whose baseline test is negative.

Secondary AIM:

1.1 To identify and describe patients with baseline UTDT positivity.

Hypothesis:

1) A subgroup of patients will demonstrate baseline positivity for UTDT. Based on previous studies, the subgroup is likely to include patients with chronic inflammatory or obstructive conditions of the pancreatic duct (pancreatic ductal adenocarcinoma, obstructive chronic pancreatitis)1 This subgroup will represent a minority (<6%) of outpatients presenting for ERCP. 1

Patients will be recruited in the pre-procedure area prior to ERCP. Only patients who would be offered ERCP as part of their previously outlined care plan will be included in this study. Patients will be screened according to inclusion/exclusion criteria described above.

Study Procedures

Informed Consent: Eligible patients will sign an IRB-approved, written informed consent to verify their willingness to participate in this study. Informed consent will be obtained on the day of their scheduled ERCP. Consent for the study will be obtained by one of the participating endoscopists and/or a research assistant. Patients will receive a copy of the signed and dated informed consent document. Original informed consent documents will be maintained on-file. A note may be made in the subject's medical record regarding participation in the research study. Once consented and enrolled into the trial, patients will be issued a unique identifier for the purposes of data entry.

Pre-Procedure data and sample collection: After obtaining informed consent, patients will be asked health questions prior to ERCP to assess and quantify current and prior alcohol use, current and prior tobacco use, quantification of narcotic use and quantification of non-steroidal anti-inflammatory drug (NSAID) use. Narcotic and NSAID use in the 7 days prior to ERCP will be recorded.

Pain scores will be collected at baseline and post ERCP. Subjects will be shown the study pain scale (appendix 1) and asked to pick a number on the scale to rate their pain at baseline and 2-3 hours (+ or - 15 minutes from time of Scope out) post ERCP.

Data will be collected on the indication of ERCP, history of acute pancreatitis, recurrent acute pancreatitis, or chronic pancreatitis, history of pancreatic surgery, presence of peri-pancreatic fluid collection and prior sphincterotomy. Prior imaging may be reviewed for the presence of pancreatic mass and/or pancreatic duct obstruction.

Baseline tests may be obtained prior to undergoing ERCP including serum pancreatic enzymes (amylase, lipase), serum liver enzymes, and coagulation profile as is the standard for our endoscopy unit. Available outpatient laboratory data within 48-72 hours of ERCP will be reviewed. Lack of baseline labs will not be a criterion for exclusion from the study.

Patients with baseline, pre-procedure positivity for UTDT (> or = 50ug/L) will undergo all study procedures as outlined below with the exception of 2 hour UTDT level.

Patients who are unable to provide a urine sample for post ERCP testing will still be included in the final analysis of baseline UTDT level. Subjects who are excluded due to the inability to access the ampulla at ERCP will also still be Included in the final analysis of baseline UTDT level.

Intra-procedural Data Collection: Patients will undergo ERCP as intended. All clinical decisions and endoscopic interventions prior to, during and after ERCP will be performed at the discretion of the treating physician. Data on duration of procedure, placement of pancreatic or biliary duct stents, ERCP maneuvers deployed for cannulation (e.g. needle knife), findings associated with chronic pancreatitis (e.g pancreatic duct stones), pancreatic duct leak, peri-procedural NSAIDs administration, amount of intraoperative IV fluids and any immediate complications including perforation, bleeding, or hemodynamic instability will be recorded.

Immediate Postoperative Care, Data and Sample collection: At our institution, patients typically remain in the recovery area for 2-3 hours after completion of the ERCP. This time interval in part is related to two-phase recovery after general anesthesia, which is the standard sedation approach for ERCP outpatients. Patients will remain for recovery after ERCP for at least two hours for a post procedure observation period and collection of UTDT result. During this time, a urine sample for UTDT testing will be collected at 2 -3 hours (+ or - 15 minutes from time of Scope out) after ERCP by the study research technician. Patients, study investigators, ERCP care team, nursing staff will be blinded to the results. The statistician will be blinded to the urine trypsinogen-2 test during statistical analysis.

The decision to admit/monitor the patient will be left to the discretion of the endoscopist / ERCP care team and will occur blinded to the UTDT results. Data regarding symptoms (e.g. nausea/vomiting, abdominal pain scores), narcotic administered for pain symptoms, duration in recovery, volume of IV fluids administered in recovery and decision to admit or discharge will be recorded.

Patients will receive a risk assessment for post-ERCP pancreatitis. This will calculated and tracked for the purposes of this study.

Follow Up Data Collection: Patients who are hospitalized will have serum amylase and lipase drawn after the ERCP procedure per standard clinical protocol timelines. Patients who are discharged to home/other after ERCP will be contacted by telephone and/or email 5 days (+ 4 days or - 2 days) and 30 days ( + or - 10 days) after the ERCP by a study team member to determine whether PEP occurred and was managed outside of our institution. Patients will be asked about ERCP procedure complications such as infection, bleeding, perforation and death. This contact may be made by phone, email or text message. Subjects will be asked for their preferred method of contact at study enrollment. Records confirming post ERCP pancreatitis will be requested if the patient is admitted and/or initially managed at an outside institution for PEP. Patients without hospitalization for symptoms attributable to post ERCP pancreatitis will be classified as not having developed PEP. Records pertaining to any ERCP procedure complications will also be requested.

PEP will be defined by the primary ERCP team. The ERCP team will be blinded to the UTDT result when determining PEP.

Clinical data regarding volume of IV fluids administered at 24, 48 hours of admission and severity of pancreatitis (based on Cotton criteria, Modified Marshall Score and graded presence of necrosis) will be assessed recorded for all patients admitted with PEP.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of Age
2. Undergoing Outpatient ERCP

Exclusion Criteria:

1. Unwillingness or inability to consent for the study
2. Acute pancreatitis on presentation or within 1 month
3. Recent ERCP (i.e. within 1 month)
4. Amylase or Lipase elevation greater than 2 x upper limit of normal within 7 days prior to ERCP
5. Stage 3 or 4 renal disease and/or oliguria
6. Inability to access the ampulla at ERCP attempt (e.g. gastric outlet obstruction)
7. Unable to provide baseline urine sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Easler, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data with other researchers

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Actim Pancreatitis Dipstick Test
Started | 394
Completed | 254
Not Completed | 140

BASELINE CHARACTERISTICS:
Population: Patients presenting for ERCP
Arm/Group | Actim Pancreatitis Dipstick Test
Number analyzed (Participants) | 254
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [45 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 157
  Male | 97
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 8
  White | 242
  More than one race | 0
  Unknown or Not Reported | 0
Indication for ERCP [Count of Participants; unit: Participants] — Some patients had overlapping indications.
  Participants
    Biliary | 167
    Pancreatic | 61
    Biliary and Pancreatic | 26
Reported Pre-ERCP abdominal pain [Count of Participants; unit: Participants] | 119
Reported Post-ERCP abdominal pain [Count of Participants; unit: Participants] — This measure is attempting to characterize participants' baseline symptoms/diagnosis. The intervention is a diagnostic urine test for post-ERCP pancreatitis, and all participants are undergoing the ERCP procedure for clinical reasons (ERCP is not a study procedure). The baseline characteristics included in the results are meant to characterize participants before the diagnostic urine test is conducted.
  Participants | 129
Post-ERCP pancreatitis [Count of Participants; unit: Participants] — This measure is attempting to characterize participants' baseline symptoms/diagnosis. The intervention is a diagnostic urine test for post-ERCP pancreatitis, and all participants are undergoing the ERCP procedure for clinical reasons (ERCP is not a study procedure). The baseline characteristics included in the results are meant to characterize participants before the diagnostic urine test is conducted.
  Participants | 9
Pre-ERCP UTDT positivity [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Urine Trypsinogen-2 Dipstick Testing for the Diagnosis of Post-ERCP Pancreatitis
Description: The urine Trypsinogen result will be codified as positive (indicative of a urine level cutpoint >50ug/L) or negative for post ERCP pancreatitis (indicative of a urine cutpoint level of <50ug/L) . This will be measured against the consensus criteria diagnosis for post ERCP pancreatitis (admission for abdominal pain symptoms of pancreatitis and serum amylase or lipase >3 times the upper limit of normal at 24 hours after ERCP).
  1. True positive: Positive dipstick, post ERCP pancreatitis diagnosis by consensus criteria
  2. True negative: negative dipstick testing, no diagnosis of post ERCP pancreatitis by consensus criteria
  3. False positive: positive urine dipstick test, no diagnosis of post-ERCP pancreatitis by consensus criteria
  4. False negative: negative urine dipstick test. diagnosis of post-ERCP pancreatitis by consensus criteria
Time Frame: Urine dipstick testing assessed 2-3 hours following ERCP, for post ERCP pancreaitits.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Actim Pancreatitis Dipstick Test
Number analyzed (Participants) | 254
percentage of participants
  Sensitivity (%) | 11.1 [7.25 to 14.98]
  Specificity (%) | 91 [87.5 to 94.54]
  Positive Predictive Value (%) | 4.4 [1.84 to 6.86]
  Negative Predictive Value | 96.5 [94.29 to 98.79]

ADVERSE EVENTS:
Time Frame: 30 days
Description: An adverse event will be consider a complication that occurred due to the collection of urine for testing or administration of health questions. Associated adverse events will be reported to the IRB per the IRB reporting criteria
Arm/Group | Actim Pancreatitis Dipstick Test
All-Cause Mortality (participants affected / at risk) | 0/394
Serious Adverse Events (participants affected / at risk) | 0/394
Other Adverse Events (participants affected / at risk) | 0/394

LIMITATIONS AND CAVEATS:
Did not meet enrollment goal for the study (goal 1825 subjects)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT03098082/Prot_SAP_000.pdf